CLINICAL TRIAL: NCT03541525
Title: Pathophysiological Explorations of Red Blood Cells
Acronym: GR-Ex
Status: Recruiting | Type: Observational
Sponsor: Imagine Institute (Other)
Responsible Party: Sponsor
Other Study IDs: IMNIS2015-04
Record Dates: First submitted 2018-03-23; First posted 2018-05-30 (Actual); Last update posted 2025-04-30 (Actual); Status verified 2025-04

CONDITIONS: Red Blood Cell Disorder

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Collection of:
  * Blood samples
  * Surgical remainders (tumor, skin, kidney,...)
  * Urine
  * Saliva
  * Hair
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Affected patients: Biological samples of blood for all patients. Biological samples of saliva, surgical remainder (skin, tumor, kidney,....), saliva, urine, hair.
  Interventions: Other: Biological sampling
- Non affected relatives: Biological samples of blood for all relatives.
  Interventions: Other: Biological sampling

INTERVENTIONS:
Other: Biological sampling — Biological samples including blood, surgical remainder, urine,...

SUMMARY:
GR-Ex is a program labelled by Labex (Laboratory of Excellence) by the French Ministry of Higher Education and Research. This program aims to develop the means to improve knowledge in the physiology and pathologies of erythropoiesis, red blood cells and iron metabolism, and to develop new therapeutic protocols capable of providing added value in terms of innovation.

ELIGIBILITY:
Inclusion Criteria:

* To be affected or have a family history of disease bound to the red blood cell,
* For adult subjects, have signed an informed consent form,
* For minor or major under legal safeguard subjects, the form must be signed by both parents (for minors) or by the legal representative,
* Be affiliated to health insurance.

Exclusion Criteria:

* Being deprived of freedom

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Inclusion of patients affected by red blood cell disorder and their non affected relatives
Sampling Method: Probability Sample
Enrollment: 3750 (Estimated)
Dates: Start 2017-10-16 (Actual); Primary Completion 2037-10-15 (Estimated); Study Completion 2037-10-15 (Estimated)

PRIMARY OUTCOMES:
Innovative markers of spleen fonctionality | 20 years
  Retention rate (%) of red blood cells using Microsphiltration compared with non affected subjects
Quantification of inflammation in sickle cell disease | 20 years
  Activation rate of circulating mastocytes (%)
Markers of post-artesunate hemolysis | 20 years
  Concentration of pitted red blood cells at day 3
Correlation between transfusion yield and the storage of red blood cell bags | 20 years
  Increasing in haemoglobin concentration at 6 hours post transfusion
Efficiency of Phosphodiesterase inhibitor on neutrophil adhesion in Sickle cell disease | 20 years
  Proportional change in adhesion rate (%) of neutrophils measured in the peripheral blood before and after treatment with phosphodiesterase inhibitors
Quantification of mitochondria removal during erythropoiesis in SDC patients, consequences on the mature RBC | 20 years
  Mitochondria rate and level of ROS in RBC measured by Flow Cytometry
Study of iron metabolism in Diamond-Blackfan Anemia patients | 20 years
  Dosage of iron metabolism parameters

CONTACTS AND LOCATIONS:
Overall Officials: Olivier Hermine, MD, PhD, Study Director — Assistance Publique - Hôpitaux de Paris
Locations (25):
- CHU Hôpital de la Mère et de l'enfant Lagune, Cotonou, Benin
- France (23):
  - CHU Amiens-Picardie, Amiens
  - Hôpital Privé d'Antony, Antony
  - Hôpital Avicenne, Bobigny
  - Hôpital Pellegrin, Bordeaux
  - Hôpital Beaujon, Clichy
  - Hôpital Louis Mourier, Colombes
  - Hopital Henri Mondor, Créteil
  - CHU Kremlin Bicetre, Le Kremlin-Bicêtre
  - Hopital de la conception, Marseille
  - Hôpital d'Enfants de la TIMONE, Marseille
  - Hôpital Saint Eloi, Montpellier
  - CHU de Niort, Niort
  - Groupe Hospitalier Diaconesses Croix Saint Simon, Paris
  - Hopital Necker - Enfants malades, Paris
  - Hôpital Armand Trousseau, Paris
  - Hôpital Cochin, Paris
  - Hôpital Européen Georges-Pompidou, Paris
  - Hôpital Robert Debré, Paris
  - Hôpital Saint Louis, Paris
  - Hôpital Saint-Antoine, Paris
  - Institut Pasteur, Paris
  - CHU de Rouen, Rouen
  - Hôpital national d'instruction des armées Bégin, Saint-Mandé
- CHU de la Guadeloupe, Pointe-à-Pitre, Guadeloupe

REFERENCES:
- [Derived] Qiang Y, Sissoko A, Liu ZL, Dong T, Zheng F, Kong F, Higgins JM, Karniadakis GE, Buffet PA, Suresh S, Dao M. Microfluidic study of retention and elimination of abnormal red blood cells by human spleen with implications for sickle cell disease. Proc Natl Acad Sci U S A. 2023 Feb 7;120(6):e2217607120. doi: 10.1073/pnas.2217607120. Epub 2023 Feb 2. PMID 36730189